CLINICAL TRIAL: NCT05292183
Title: Neuromodulation of Affective Valence in Humans by Amygdala Stimulation
Brief Title: Modulation of Emotion Perception in Humans Via Amygdala Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Krzysztof Bujarski, Section Chief, Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY02001399; 1R21MH124674-01A1 (NIH)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Refractory Epilepsy
Keywords: Human Amygdala; Deep Brain Stimulation; Psychiatric Disorders
MeSH Terms: conditions — Drug Resistant Epilepsy; Mental Disorders | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: The researchers will use computerized randomization of electrical stimulation for each participant. The stimulation vs non stimulation are not discrete events and occur in random order within individual participants during each daily testing session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stimulation (Experimental): This part will include 24 randomly chosen images from each of four categories (total of 96 images varying in valence and arousal) and will be presented block-randomized amygdala stimulation.
  Interventions: Other: Electrical Stimulation
- No stimulation (No Intervention): This part will include 24 randomly chosen images from each of four categories (total of 96 images varying in valence and arousal) and will be presented without amygdala stimulation.

INTERVENTIONS:
Other: Electrical Stimulation — We will use a computer randomized stimulation of specific areas in the amygdala while showing a computer randomized set of pictures.
  Arms: Stimulation

SUMMARY:
This study will enroll patients with epilepsy who are being evaluated for epilepsy surgery and have intracranial EEG electrodes. In this study, the aim is to record brain signals from areas important in social and emotional processing and to understand how electrical brain stimulation - called neuromodulation - affects such processing. Patients enrolled in this study will be asked to view images depicting a variety of emotionally positive, negative, or neutral themes. As the patient views these images, a small amount of imperceptible and painless electric current will be used to map function of certain parts of a human brain. The overarching goal of the study is to determine if neuromodulation can be used in certain areas of the brain to treat cognitive disorders such as memory loss and post-traumatic stress disorder.

DETAILED DESCRIPTION:
One to two study tasks will be performed by each participant to help us understand how the brain processes emotion and how stimulation effects emotional processing.

These study tasks will last up to several minutes each, and generally require participants to view pictures while EEG recordings are made from the electrodes placed in specific areas of the brain. The routine video/EEG monitoring and brain function testing should not be disrupted or prolonged by the study testing, and if a participant has a seizure during the testing, it will be recorded as usual for review by participant's providers.

The following study procedures will likely be carried out in each individual case:

1. Recording from areas important in social and emotional processing.

   A computer monitor will be used to present pictures of people engaged in social interaction. Additionally, the researchers will present individual participants with well standardized tasks designed to understand the nature of emotions. Some of these images may be emotionally disturbing. Should participants become uncomfortable with viewing such images, participants would be provided with a choice to not participate in this study.
2. Using brain stimulation to map function of certain parts of your brain.

   A brain stimulator will be used -normally used to map where important brain regions are located-to understand new functions of the brain. Each participant will be presented with pictures on a computer screen. As participant(s) views these pictures, the brain stimulator may be activated (this is not something that is felt by a person) and an electrical stimulation through the implanted electrodes will be delivered to specific regions of the brain. Research team will be measuring how brain stimulation may affect each individual's emotional response to a specific stimulus.
3. Completing the Emotion Self-Rating (ESR) Scale.

This questionnaire will be given to ensure the stimulation doesn't increase any unpleasant emotional experience for participants. This will take place before and during the stimulation of a specific part of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* FSIQ 75 and above or any equivalent test of generalized intelligence as determined by the PI to adequately predict engagement in the task
* Able to give independent consent for participation in the study

Exclusion Criteria:

* Additional neurological disorders (such as dementia, stroke, brain tumor, etc.)
* Any psychiatric condition that would limit their ability to provide consent and/or perform study tasks within normal limits. This would be based on presurgical psychiatric assessment.
* Anything else, that in the opinion of the principal investigator, might preclude them from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof A Bujarski, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
The study results will be available on ClinicalTrials.gov and will be published in appropriate clinical journal upon completion.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 15 patients who completed the study, EEG data was of adequate quality for analysis for four (4) patients, behavioral data with amygdala stimulation was available for nine (9) patients.
Groups:
- Entire Study Population: This is the group that was recruited and were able to complete testing
Period: Overall Study
Arm/Group | Entire Study Population
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: This population is the same as the recruited patients in participant flow
Groups:
- The Entire Study Population: This part will include 24 randomly chosen images from each of four categories (total of 96 images varying in valence and arousal) and will be presented block-randomized amygdala stimulation and no stimulation. All participants received sham and actual stimulation, however, the order in which the stimuli (with or without stimulation) were presented to the participants was computer randomized. The order in which the stimuli were presented was unique to each individual participant
  Electrical Stimulation: We will use a computer randomized stimulation of specific areas in the amygdala while showing a computer randomized set of pictures.
  No Electrical stimulation: we will use a computer randomized sham stimulation of specific areas in the amygdala while showing a computer randomized set of pictures
Arm/Group | The Entire Study Population
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Z-score Gamma Power in Amygdala Per Valence Category
Description: Valence of each image is assessed by each subject using a Likert-type rating scale with a range of 1 to 7, where 1 represents most negative valence, 4 as neutral, and 7 as most positive. Valence categories are defined in the following manner: negative = 1.0 to 3.0, neutral = 3.1 to 5.0, negative = 5.1 to 7.0. Activation is measured by gamma frequency power (mµV²/30-100 Hz) at 0-1000 msec following image presentation in the basolateral amygdala electrode contact and compared to baseline defined as -500 msec to 0 of image presentation. Gamma power is transformed to z-score (baseline to following image presentation) for individual observations. Z-score of 0 indicates no change from baseline. Positive z-score indicates activation of the basolateral amygdala compared to baseline. Gamma frequency range is defined as 30-100 Hz in intracranial EEG. Power was estimated via a multitaper time-frequency transformation approach. Statistics was done using linear-mixed effects models (LMEs).
Time Frame: 0 to 1000 MS following image presentation
Population: Electrophysiological data is available in 4 participants.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Gamma Power in the Amygdala According to Valence Category: This measure reflects changes in the activation of the amygdala when viewing images of specific emotional valence across all subjects. In our study, activation on intracranial EEG is measured by change in the power of the gamma band. This band is defined as frequency ranges from 30-100 Hz in intracranial EEG. An increase in gamma power reflects increased local neuronal activity during the cognitive process in question. Here we present neutral, positive, and negative valence images and determine change in gamma power for each valence category. Significant changes in gamma power from baseline is measured as z-score compared to baseline.
Arm/Group | Gamma Power in the Amygdala According to Valence Category
Number analyzed (Participants) | 4
z-score
  Gamma power positive images | 1.21 (0.23)
  Gamma power, negative valence images | 1.88 (0.78)
  Gamma power, neutral images | 1.24 (0.24)

2. Primary Outcome: Effect of Amygdala Stimulation on Perception of Valence
Description: Here we assess the effect of basolateral amygdala stimulation on valence ratings. Participants rate the emotional valence of each image in a Likert scale range of 1-7 (1= maximum negative valence, 4=maximum neutral valence, and 7 maximum positive valence) for each of the 96 images. We randomly apply electrical stimulation during perception and of 50% of the images presented. We analyze the effect of stimulation on image rating in the following manner: we grouped the images into three categories, negative (1 to 3), neutral (3.1 to 5), and positive (5.1 to 7) based on subject specific ratings. 2. We then used a multivariate model to assess the effect of stimulation on perception of neutral, negative, and positive categories across 9 patients.
Time Frame: Valence ratings were assessed immediately following the viewing of each image during performance of the task.
Population: These patients represent recruited patients that underwent stimulation of the amygdala during viewing of images of different valence.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Entire Study Population: This part will include 24 randomly chosen images from each of four categories (total of 96 images varying in valence and arousal) and will be presented block-randomized amygdala stimulation and no stimulation.
  Electrical Stimulation: We will use a computer randomized stimulation of specific areas in the amygdala while showing a computer randomized set of pictures
  No electrical stimulation:
  This includes all participants consented to be in this study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 9
units on a scale
  Neutral no stimulation | 3.27 (0.78)
  Neutral stimulation | 3.64 (0.48)
  Positive valence; no stimulation | 5.26 (0.67)
  Positive valence; stimulation | 5.08 (0.94)
  Negative valence, no stimulation | 2.02 (0.66)
  Negative valence, stimulation | 2.08 (0.59)

ADVERSE EVENTS:
Time Frame: during testing sessions for this study or 1 day
Arm/Group | Stimulation | No Stimulation
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation (N=15) | No Stimulation (N=15)
Covid-19 Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT05292183/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT05292183/ICF_001.pdf